CLINICAL TRIAL: NCT01854645
Title: A Randomized, Double Blind, Chronic Dosing, Placebo-Controlled, Parallel Group, Multi Center Study to Assess the Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe COPD, Compared With Placebo and Spiriva® Handihaler® (Tiotropium Bromide 18 µg Open-Label) as an Active Control
Brief Title: Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD); (PINNACLE 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003006-00
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- GFF MDI (Experimental): Glycopyrronium Formoterol Fumarate (GFF) Metered Dose Inhaler (MDI) (PT003)
  Interventions: Drug: GFF MDI
- GP MDI (Experimental): Glycopyrronium (GP) MDI (PT001)
  Interventions: Drug: GP MDI
- FF MDI (Experimental): Formoterol Fumarate (FF) MDI (PT005)
  Interventions: Drug: FF MDI
- Open-label tiotropium bromide inhalation powder (Active Comparator): Open-label tiotropium bromide inhalation powder (Spiriva® Handihaler®)
  Interventions: Drug: Open-label tiotropium bromide inhalation powder (Spiriva® Handihaler®)
- Placebo (Placebo Comparator): Placebo MDI
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: GFF MDI — GFF MDI administered as two puffs Bis in Di.e. Twice Daily (BID)
  Arms: GFF MDI
Drug: GP MDI — GP MDI administered as two puffs BID
  Arms: GP MDI
Drug: FF MDI — FF MDI administered as two puffs BID
  Arms: FF MDI
Drug: Open-label tiotropium bromide inhalation powder (Spiriva® Handihaler®) — Taken as 1 capsule daily containing 18 µg of open-label tiotropium via the Handihaler dry powder inhaler (DPI)
  Arms: Open-label tiotropium bromide inhalation powder
Drug: Placebo MDI — Inhaled placebo administered as two puffs BID
  Arms: Placebo

SUMMARY:
The overall objective of this study is to assess the efficacy and safety of treatment with PT003 (GFF MDI), PT005 (FF MDI), PT001 (GP MDI), and open-label tiotropium bromide inhalation powder compared with each other and Placebo MDI over 24 weeks in subjects with moderate to very severe COPD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects at least 40 years of age and no older than 80 at Visit 1.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Average f the -60 and the -30 min pre-dose FEV1 assessments must be < 80% predicted normal value calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations.
* Subjects willing and, in the opinion of the investigator, able to adjust current COPD therapy as required by the protocol

Key Exclusion Criteria:

* Significant diseases other than COPD, i.e. disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Current diagnosis of asthma or alpha-1 antitrypsin deficiency
* Other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnea
* Hospitalized due to poorly controlled COPD within 3 months prior to screening or during the Screening Period
* Poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to screening or during the Screening Period
* Lower respiratory tract infections that required antibiotics within 6 weeks prior to screening or during the Screening Period
* Unstable ischemic heart disease, left ventricular failure, or documented myocardial infarction within 12 months of enrollment.
* Recent history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft within the past three months
* Congestive heart failure (CHF) New York Heart Association (NYHA) Class III/IV)
* Clinically significant abnormal 12-lead ECG
* Abnormal liver function tests defined as aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin ≥ 1.5 times upper limit of normal at Visit 1 and on repeat testing
* Cancer not in complete remission for at least five years
* History of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, lactose/milk protein or any component of the MDI

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2103 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Director — Pearl Therapeutics, Inc.
Locations (139):
- United States (121):
  - Pearl Investigative Site, Andalusia, Alabama
  - Pearl Investigative Site, Anniston, Alabama
  - Pearl Investigative Site, Athens, Alabama
  - Pearl Investigative Site, Birmingham, Alabama
  - Pearl Investigative Site, Mesa, Arizona
  - Pearl Investigative Site, Phoenix, Arizona
  - Pearl Investigative Site, Scottsdale, Arizona
  - Pearl Investigative Site, Tucson, Arizona
  - Pearl Investigative Site, Anaheim, California
  - Pearl Investigative Site, Carlsbad, California
  - Pearl Investigative Site, Lakewood, California
  - Pearl Investigative Site, Los Angeles, California
  - Pearl Investigative Site, Pasadena, California
  - Pearl Investigative Site, Poway, California
  - Pearl Investigative Site, Sacramento, California
  - Pearl Investigative Site, San Diego, California
  - Pearl Investigative Site, Tustin, California
  - Pearl Investigative Site, Vista, California
  - Pearl Investigative Site, Colorado Springs, Colorado
  - Pearl Investigative Site, Denver, Colorado
  - Pearl Investigative Site, Fort Collins, Colorado
  - Pearl Investigative Site, Wheat Ridge, Colorado
  - Pearl Investigative Site, Danbury, Connecticut
  - Pearl Investigative Site, Waterbury, Connecticut
  - Pearl Investigative Site, Brandon, Florida
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Lehigh Acres, Florida
  - Pearl Investigative Site, Miami, Florida
  - Pearl Investigative Site, Ormond Beach, Florida
  - Pearl Investigative Site, Panama City, Florida
  - Pearl Investigative Site, Pensacola, Florida
  - Pearl Investigative Site, St. Petersburg, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Atlanta, Georgia
  - Pearl Investigative Site, Austell, Georgia
  - Pearl Investigative Site, Columbus, Georgia
  - Pearl Investigative Site, Duluth, Georgia
  - Pearl Investigative Site, Gainesville, Georgia
  - Pearl Investigative Site, Coeur d'Alene, Idaho
  - Pearl Investigative Site, Champaign, Illinois
  - Pearl Investigative Site, Evanston, Illinois
  - Pearl Investigative Site, Peoria, Illinois
  - Pearl Investigative Site, River Forest, Illinois
  - Pearl Investigative Site, Anderson, Indiana
  - Pearl Investigative Site, Avon, Indiana
  - Pearl Investigative Site, Elwood, Indiana
  - Pearl Investigative Site, Evansville, Indiana
  - Pearl Investigative Site, Iowa City, Iowa
  - Pearl Investigative Site, Topeka, Kansas
  - Pearl Investigative Site, Louisville, Kentucky
  - Pearl Investigative Site, Lafayette, Louisiana
  - Pearl Investigative Site, Sunset, Louisiana
  - Pearl Investigative Site, Baltimore, Maryland
  - Pearl Investigative Site, Hollywood, Maryland
  - Pearl Investigative Site, Livonia, Michigan
  - Pearl Investigative Site, Southfield, Michigan
  - Pearl Investigative Site, Edina, Minnesota
  - Pearl Investigative Site, Fridley, Minnesota
  - Pearl Investigative Site, Minneapolis, Minnesota
  - Pearl Investigative Site, Woodbury, Minnesota
  - Pearl Investigative Site, Saint Charles, Missouri
  - Pearl Investigative Site, Springfield, Missouri
  - Pearl Investigative Site, St Louis, Missouri
  - Pearl Investigative Site, Missoula, Montana
  - Pearl Investigative Site, Bellevue, Nebraska
  - Pearl Investigative Site, Omaha, Nebraska
  - Pearl Investigative Site, Las Vegas, Nevada
  - Pearl Investigative Site, Ocean City, New Jersey
  - Pearl Investigative Site, Albuquerque, New Mexico
  - Pearl Investigative Site, Corning, New York
  - Pearl Investigative Site, Burlington, North Carolina
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Greensboro, North Carolina
  - Pearl Investigative Site, Huntersville, North Carolina
  - Pearl Investigative Site, Raleigh, North Carolina
  - Pearl Investigative Site, Wilmington, North Carolina
  - Pearl Investigative Site, Winston-Salem, North Carolina
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Columbus, Ohio
  - Pearl Investigative Site, Dayton, Ohio
  - Pearl Investigative Site, Dublin, Ohio
  - Pearl Investigative Site, Oregon, Ohio
  - Pearl Investigative Site, Bend, Oregon
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Portland, Oregon
  - Pearl Investigative Site, Monroeville, Pennsylvania
  - Pearl Investigative Site, Philadelphia, Pennsylvania
  - Pearl Investigative Site, Charleston, South Carolina
  - Pearl Investigative Site, Easley, South Carolina
  - Pearl Investigative Site, Gaffney, South Carolina
  - Pearl Investigative Site, Greenville, South Carolina
  - Pearl Investigative Site, Mt. Pleasant, South Carolina
  - Pearl Investigative Site, Murrells Inlet, South Carolina
  - Pearl Investigative Site, Myrtle Beach, South Carolina
  - Pearl Investigative Site, Rock Hill, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, Union, South Carolina
  - Pearl Investigative Site, Rapid City, South Dakota
  - Pearl Investigative Site, Bristol, Tennessee
  - Pearl Investigative Site, Johnson City, Tennessee
  - Pearl Investigative Site, Kingsport, Tennessee
  - Pearl Investigative Site, Tullahoma, Tennessee
  - Pearl Investigative Site, Austin, Texas
  - Pearl Investigative Site, El Paso, Texas
  - Pearl Investigative Site, Fort Worth, Texas
  - Pearl Investigative Site, Houston, Texas
  - Pearl Investigative Site, Huntsville, Texas
  - Pearl Investigative Site, Longview, Texas
  - Pearl Investigative Site, Lufkin, Texas
  - Pearl Investigative Site, New Braunfels, Texas
  - Pearl Investigative Site, San Antonio, Texas
  - Pearl Investigative Site, Midvale, Utah
  - Pearl Investigative Site, Salt Lake City, Utah
  - Pearl Investigative Site, South Burlington, Vermont
  - Pearl Investigative Site, Abingdon, Virginia
  - Pearl Investigative Site, Richmond, Virginia
  - Pearl Investigative Site, Spokane, Washington
  - Pearl Investigative Site, Tacoma, Washington
  - Pearl Investigative Site, Morgantown, West Virginia
  - Pearl Investigative Site, West Allis, Wisconsin
- Australia (12):
  - Pearl Investigative Site, New Lambton, New South Wales
  - Pearl Investigative Site, Westmead, New South Wales
  - Pearl Investigative Site, Brisbane, Queensland
  - Pearl Investigative Site, Cairns, Queensland
  - Pearl Investigative Site, Wooloongabba, Queensland
  - Pearl Investigative Site, Adelaide, South Australia
  - Pearl Investigative Site, Daw Park, South Australia
  - Pearl Investigative Site, Toorak Gardens, South Australia
  - Pearl Investigative Site, Box Hill, Victoria
  - Pearl Investigative Site, Heidelberg, Victoria
  - Pearl Investigative Site, Nedlands, Western Australia
  - Pearl Investigative Site, Perth, Western Australia
- New Zealand (6):
  - Pearl Investigative Site, Otahuhu, Aukland
  - Pearl Investigative Site, Caversham, Dunedin
  - Pearl Investigative Site, Greenlane, East Aukland
  - Pearl Investigative Site, Hamilton, Waikato Region
  - Pearl Investigative Site, Newtown, Wellington Region
  - Pearl Investigative Site, Tauranga

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Martinez FJ, Lipworth BJ, Rabe KF, Collier DJ, Ferguson GT, Sethi S, Feldman GJ, O'Brien G, Jenkins M, Reisner C. Benefits of glycopyrrolate/formoterol fumarate metered dose inhaler (GFF MDI) in improving lung function and reducing exacerbations in patients with moderate-to-very severe COPD: a pooled analysis of the PINNACLE studies. Respir Res. 2020 May 25;21(1):128. doi: 10.1186/s12931-020-01388-y. PMID 32450869
- [Derived] Martinez FJ, Rabe KF, Lipworth BJ, Arora S, Jenkins M, Martin UJ, Reisner C. Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Improves Lung Function versus Monotherapies in GOLD Category A Patients with COPD: Pooled Data from the Phase III PINNACLE Studies. Int J Chron Obstruct Pulmon Dis. 2020 Jan 9;15:99-106. doi: 10.2147/COPD.S229794. eCollection 2020. PMID 32021148
- [Derived] Martinez FJ, Fabbri LM, Ferguson GT, Orevillo C, Darken P, Martin UJ, Reisner C. Baseline Symptom Score Impact on Benefits of Glycopyrrolate/Formoterol Metered Dose Inhaler in COPD. Chest. 2017 Dec;152(6):1169-1178. doi: 10.1016/j.chest.2017.07.007. Epub 2017 Jul 16. PMID 28720336
- See also: PT003006-02 Protocol and Amendment-FINAL-Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4154&filename=PT003006-02%20Protocol%20Amendment-FINAL-11Sept14_29Jun16_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 160 sites throughout the US, Australia, and New Zealand from June 2013 - February 2015. Study participation was a maximum of 32 weeks.
Pre-assignment Details: Study was a multicenter, randomized, double-blind, parallel group, chronic dosing, active- and placebo-controlled study; each patient was randomized to receive 1 of 5 possible treatments over the course of a 24-week treatment period
Groups:
- GFF MDI (PT003): Glycopyrronium Formoterol Fumarate (GFF) Metered Dose Inhaler (MDI) 14.4/9.6 mcg
- GP MDI (PT001): Glycopyrronium (GP) MDI 14.4 mcg
- FF MDI (PT005): Formoterol Fumarate (FF) MDI 9.6 mcg
- Spiriva® Handihaler® (Open-label): Open-label tiotropium bromide inhalation powder 18 mcg
Period: Overall Study
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Started | 527 | 451 | 452 | 453 | 220
Completed | 429 | 345 | 370 | 391 | 160
Not Completed | 98 | 106 | 82 | 62 | 60
Not completed — Protocol-Specified Criteria | 13 | 10 | 8 | 5 | 7
Not completed — Administrative Reasons / Missing | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 0 | 5 | 4 | 1
Not completed — Lost to Follow-up | 10 | 7 | 8 | 5 | 0
Not completed — Physician Decision | 1 | 5 | 3 | 3 | 7
Not completed — Withdrawal by Subject | 31 | 41 | 30 | 21 | 24
Not completed — Lack of Efficacy | 7 | 12 | 9 | 3 | 9
Not completed — Adverse Event | 33 | 31 | 19 | 20 | 11

BASELINE CHARACTERISTICS:
Population: 7 subjects were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo | Total
Number analyzed (Participants) | 526 | 451 | 449 | 451 | 219 | 2096
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (8.4) | 62.9 (8.4) | 63.0 (8.3) | 63.0 (8.6) | 62.5 (8.3) | 62.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 196 | 203 | 182 | 97 | 914
  Male | 290 | 255 | 246 | 269 | 122 | 1182

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 24
Description: Change from baseline in morning pre-dose trough forced expiratory volume in 1 second (FEV1) at Week 24
Time Frame: Baseline and at Week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 429 | 344 | 367 | 390 | 161
Liters | 0.126 [0.107 to 0.145] | 0.066 [0.045 to 0.087] | 0.062 [0.041 to 0.082] | 0.105 [0.084 to 0.125] | -0.024 [-0.055 to 0.007]

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 Over 24 Weeks
Description: Change from baseline in morning pre-dose trough forced expiratory volume in 1 second (FEV1) over 24 weeks. FEV1 was assessed at multiple time points post-baseline,and a modelbased average of all visits starting from Week 2 through week 24 inclusive was calculated. The change values reported in the table represent the change between the baseline and the average FEV1 post-baseline.
Time Frame: Baseline and Weeks 2 to 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 519 | 440 | 439 | 446 | 208
Liters | 0.150 [0.136 to 0.164] | 0.091 [0.076 to 0.106] | 0.086 [0.071 to 0.101] | 0.122 [0.107 to 0.137] | -0.007 [-0.029 to 0.015]

3. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Score
Description: Change from baseline in the SGRQ total score. The SGRQ is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of GFF MDI, FF MDI and GP MDI on health-related quality of life as compared to placebo in subjects with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life.
Time Frame: Baseline and at Week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 503 | 425 | 434 | 435 | 213
Scores on a scale | -3.1 [-4.0 to -2.2] | -1.2 [-2.2 to -0.2] | -2.4 [-3.4 to -1.4] | -2.7 [-3.6 to -1.7] | -0.8 [-2.2 to 0.7]

4. Secondary Outcome: Rescue Ventolin Hydrofluoroalkane (HFA) Use
Description: Change from baseline in average daily rescue Ventolin HFA use
Time Frame: Baseline and at Week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs / Day
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 525 | 449 | 446 | 449 | 218
Puffs / Day | -0.8 [-1.0 to -0.6] | -0.5 [-0.7 to -0.3] | -0.8 [-1.0 to -0.6] | -0.4 [-0.6 to -0.2] | 0.3 [0.0 to 0.6]

5. Secondary Outcome: Onset of Action as Assessed by FEV1
Description: Defined as the first time-point using the 5- and 15-minute post dose measurements where the difference in FEV1 from Placebo was statistically significant
Time Frame: Assessed for 5- and 15-minute post dose on Day 1
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 418 | 363 | 366 | 364 | 172
Liters
  5 min post dose | 0.185 [0.175 to 0.195] | 0.042 [0.031 to 0.053] | 0.182 [0.171 to 0.193] | 0.048 [0.037 to 0.059] | -0.002 [-0.017 to 0.014]
  15 min post dose | 0.226 [0.216 to 0.237] | 0.101 [0.090 to 0.113] | 0.212 [0.201 to 0.224] | 0.117 [0.105 to 0.129] | 0.022 [0.005 to 0.038]
Statistical Analysis 1: Comparison: GFF MDI (PT003) vs Placebo; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: GFF MDI (PT003) vs Placebo; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: GP MDI (PT001) vs Placebo; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: GP MDI (PT001) vs Placebo; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: FF MDI (PT005) vs Placebo; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 6: Comparison: FF MDI (PT005) vs Placebo; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA

6. Secondary Outcome: Peak Change From Baseline in FEV1 Within 2 Hours Post-dose
Description: Peak change from baseline in forced expiratory volume in 1 second (FEV1) within 2 hours post-dose
Time Frame: Baseline and at Week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Number analyzed (Participants) | 428 | 343 | 367 | 388 | 160
Liters | 0.356 [0.335 to 0.377] | 0.223 [0.200 to 0.246] | 0.263 [0.240 to 0.285] | 0.259 [0.237 to 0.281] | 0.065 [0.031 to 0.098]

ADVERSE EVENTS:
Time Frame: SAEs and AEs were collected throughout study participation and for two weeks after study completion.
Description: Safety population included all participants who received at least one dose of investigational drug participants were included in safety population according to the investigational drug received
Arm/Group | GFF MDI (PT003) | GP MDI (PT001) | FF MDI (PT005) | Spiriva® Handihaler® (Open-label) | Placebo
Serious Adverse Events (participants affected / at risk) | 44/526 | 36/451 | 29/452 | 36/451 | 16/220
Other Adverse Events (participants affected / at risk) | 73/526 | 59/451 | 57/452 | 58/451 | 47/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GFF MDI (PT003) (N=526) | GP MDI (PT001) (N=451) | FF MDI (PT005) (N=452) | Spiriva® Handihaler® (Open-label) (N=451) | Placebo (N=220)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 17 (20) | 8 (8) | 8 (8) | 7 (7)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistatxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 7 (7) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lobar pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Opthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Translational cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Inflamation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0/1 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) (N=526) | GP MDI (PT001) (N=451) | FF MDI (PT005) (N=452) | Spiriva® Handihaler® (Open-label) (N=451) | Placebo (N=220)
Nasopharyngitis (Infections and infestations) | 43 (45) | 23 (24) | 28 (32) | 26 (26) | 18 (21)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 20 (21) | 14 (14) | 17 (18) | 16 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 16 (19) | 15 (16) | 15 (15) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.